CLINICAL TRIAL: NCT00220155
Title: A Phase II Trial of Fixed Dose Rate Gemcitabine in Patients With Advanced or Metastatic Colorectal Cancer.
Brief Title: Phase II Fixed Dose Rate Gemcitabine for Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2398
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemcitabine

SUMMARY:
To assess the efficacy and safety of gemcitabine given by fixed dose rate intravenous infusion in patients with pretreated metastatic colorectal cancer.

DETAILED DESCRIPTION:
Previous lines of treatment recorded. Adjuvant and palliative.

Treatment will continue until clinical indication due to PD or toxicity, or until completion of 6 cycles of gemcitabine, whichever comes first.

All patients will be assessed for toxicity and followed up for disease recurrence/progression.

The study will be divided into two accrual stages - the first consisting of 17 patients. If 6 or more patients achieve tumour response or stabilisation in the first stage, the second stage will commence accrual of a further 20 patients. Hence, the total planned accrual will be 37 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histologically proven colorectal adenocarcinoma.
* Locally advanced (inoperable) or metastatic colorectal carcinoma treated with at least one prior chemotherapy regimen.
* Progressive disease documented by CT either during or within 3 months of completion of previous chemotherapy
* No previous malignant disease other than non-melanotic skin cancer or carcinoma-in-situ of the uterine cervix.
* Unidimensional measurable disease as assessed by CT.
* Adequate bone marrow function; Hb >10g/dl, platelets >100 x109/l, WBC >3x109/l, Neut >1.5x109/l.
* Adequate liver function: Serum Bilirubin <1.5 x upper limit of normal
* Adequate renal function: Serum Creatinine < 0.11 mmol/L
* No concurrent uncontrolled medical conditions
* WHO performance status 0,1 or 2
* Adequate contraceptive precautions, if appropriate
* Informed written consent
* Negative pregnancy test in women of child bearing age
* Life expectancy > 3 months

Exclusion Criteria:

* Medical or psychiatric condition that comprise the patient's ability to take informed consent.
* Patients within 4 weeks of chemotherapy or radiotherapy (6 weeks for nitrosureas or mitomycin C).
* Previous treatment with gemcitabine.
* Patients with uncontrolled cerebral metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-05

PRIMARY OUTCOMES:
Proportion of patients obtaining disease control in the form of tumour response or stabilisation

SECONDARY OUTCOMES:
Treatment related toxicity
Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom